CLINICAL TRIAL: NCT05711654
Title: The Effect of Health Coaching on Perceived Social Support in Patients With Chronic Obstructive Pulmonary Disease: A Randomized Controlled Study
Brief Title: Chronic Obstructive Pulmonary Disease and Health Coaching
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harran University (Other)
Collaborators: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Derya TÜLÜCE, Faculty of Health Sciences, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Osmaniye Korkut Ata University
Record Dates: First submitted 2023-01-16; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Health coaching; Social support; Symptom management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Factorial Assignment
Who Masked: Participant
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health coaching group (Experimental): The patients in the health coaching group will first be given data collection tools, and then the COPD patient information training created by the researcher will be given.
  For the first eight weeks after the training, face-to-face meetings will be held with patients once a week.
  Data collection tools will be applied to the patients again in the fourth week and 12 weeks after the interviews are over.
  Interventions: Behavioral: Health coaching
- Control group (No Intervention): Data collection tools will be applied to the patients in the control group first, and then the COPD patient information training created by the researcher will be given.
  After the training, there will be no interviews with the patients, and data collection tools will be applied again in the 12th and 20th weeks.

INTERVENTIONS:
Behavioral: Health coaching — Coaching interview will be held with patients at regular intervals.
  Arms: Health coaching group

SUMMARY:
The aim of this study is to determine the effect of the health coaching approach applied to patients with Chronic Obstructive Pulmonary Disease on the perceived social support of the patients.

Research Hypotheses:

H0: Health coaching approach has no effect on perceived social support in patients with COPD.

H1: Health coaching approach has an effect on perceived social support in patients with COPD.

DETAILED DESCRIPTION:
The current study is in the design of a single-blind randomized controlled trial. Patients were randomized into intervention group (n:34) and control group (n=34). Coaching interview will be held once a week for 6-8 weeks with the patients in the coaching group. Coaching sessions will be based on the social support the patient receives from family and friends.

Both the coaching group and the control group will be given information about COPD. This information will be given face to face first. Later, the booklet of the training given will be delivered to the patients via message.

The data was collected using the socio-demographic information form,COPD Assessment Test (CAT), and Multidimensional Scale of Perceived Social Support (MSPSS).

Data Analysis will be done with SPSS package program

ELIGIBILITY:
Inclusion Criteria:

* over 40 years old,
* diagnosed with COPD for at least 6 months,
* without stage III and IV heart failure,
* without any cancer diagnosis,
* no communication problems (such as those who do not have problems in expressing - themselves, no hearing problems),
* not diagnosed with cognitive and mental dysfunction (such as Alzheimer's, dementia, bipolar disorder, major depression)
* Patients who agree to participate in the study will be formed.

Exclusion Criteria:

* with any cancer
* with stage IV heart failure
* patients requiring clinical follow-up due to acute COPD exacerbation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Social support | A 6-8 week coaching interview will be held with each patient participating in the study. Each patient will be followed for a total of 20 weeks.
  The social support levels perceived by the patients will be measured.The scale developed by Zimmet, Dahlem, Zimet, and Farley (1988) was adapted to Turkish by Eker et al. (2001) via its application to 50 psychiatry patients, 50 surgery patients and 50 normal individuals. The average participant age was 36. Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item scale with three sub-factors such as family, friends and significant other. Each sub-factor consists of four items. The scale is a 7-point Likert type including choices ranging from very strongly disagree (1) to very strongly agree (7). Higher scores obtained from the scale point to high levels of perceived social support.

SECONDARY OUTCOMES:
symptom managament | A 6-8 week coaching interview will be held with each patient participating in the study. Each patient will be followed for a total of 20 weeks.
  Symptoms of Patients with COPD will be measured. The CAT was used to assess symptom burden in this study. The CAT, a patient-reported scale, evaluates the effect of COPD symptoms on an individual's health. The scale consists of eight items including cough, phlegm, chest tightness, breathlessness, activities, confidence, sleep and energy. Each item is rated on a six-point Likert scale ranging from 0 (no symptom) to 5 (very serious). The total score ranges from 0 to 40 points, with lower scores indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Derya Tülüce, PhD, Principal Investigator — Osmaniye Korkut Ata University
Locations (1):
- Osmaniye Korkut Ata University, Osmaniye, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No